CLINICAL TRIAL: NCT02515058
Title: Ridge Preservation Following Tooth Extraction Using Mineralized Freeze-Dried Bone Allograft Compared to PUROS Mineralized Bone Allograft
Brief Title: Ridge Preservation Following Tooth Extraction Using Two Mineralized Cancellous Bone Allografts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Brian L Mealey, Professor and Graduate Program Director, Periodontics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0552H
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-11

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PUROS (Non-Freeze-Dried bone allograft) (Experimental): Ridge preservation bone grafting surgery with Non-Freeze-Dried cancellous bone allograft (PUROS)
  Interventions: Device: PUROS (Ridge Preservation bone grafting surgery)
- FDBA (Freeze-Dried bone allograft) (Active Comparator): Ridge preservation bone grafting surgery with Freeze-Dried cancellous bone allograft (FDBA)
  Interventions: Device: FDBA (Ridge Preservation bone grafting surgery)

INTERVENTIONS:
Device: PUROS (Ridge Preservation bone grafting surgery) — Ridge preservation bone grafting after tooth extraction
  Arms: PUROS (Non-Freeze-Dried bone allograft)
Device: FDBA (Ridge Preservation bone grafting surgery) — Ridge preservation bone grafting after tooth extraction
  Arms: FDBA (Freeze-Dried bone allograft)

SUMMARY:
The study is a 2-arm, parallel-design, randomized, prospective clinical trial designed to examine histologic wound healing following ridge preservation using bone allograft that has been prepared by either freeze-drying or via a non-freeze-dried solvent process.This entire protocol involves procedures that are standard care. All materials are FDA-approved materials being used in an FDA-approved manner. The test group subjects will have extraction sockets grafted with a cancellous non-freeze-dried bone allograft (called PUROS graft). This test group will be compared to an active control group using cancellous freeze-dried bone allograft (called FDBA). The null hypothesis is that there will be no significant difference in formation of new vital bone between treatment groups (primary outcome).

Each subject will provide a single non-molar tooth site for study treatment. After tooth extraction, the graft material will be placed and covered by a resorbable collagen membrane. Following 3 months of healing, the dental implant will be place, at which time a core of bone will be removed from the site as part of the preparation for the implant. The core biopsy will then be evaluated for the primary histologic outcome of % vital bone formation and secondary histologic outcome of % residual graft material.

DETAILED DESCRIPTION:
The study is designed to examine histologic wound healing following ridge preservation using cancellous bone allograft that has been prepared either by freeze-drying (FDBA) or by a solvent-based processing method (PUROS). This entire protocol involves procedures that are standard care. All materials are FDA-approved materials being used in an FDA-approved manner. The test group subjects will have extraction sockets grafted with a cancellous non-freeze-dried bone allograft (called PUROS graft). This test group will be compared to an active control group using cancellous freeze-dried bone allograft (called FDBA). The null hypothesis is that there will be no significant difference in formation of new vital bone between treatment groups (primary outcome).

Each subject will provide a single non-molar tooth site for study treatment. After tooth extraction, the graft material will be placed and covered by a resorbable collagen membrane. Following 3 months of healing, the dental implant will be place, at which time a core of bone will be removed from the site as part of the preparation for the implant. The core biopsy will then be evaluated for the primary histologic outcome of % vital bone formation and secondary histologic outcome of % residual graft material.

ELIGIBILITY:
Inclusion Criteria:Patients will be included in this study if they qualify the following inclusion criteria:

* Live within 50 miles from the School of Dentistry, University of Texas Health Science Center at San Antonio
* Are able to attend a minimum of 6 visits over a 4-5 month period, as required by the study protocol
* A single rooted tooth that has been identified as requiring extraction
* Desire a dental implant to replace the missing tooth
* Have adequate restorative space for a dental implant-retained restoration
* Have at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.
* Have a dehiscence of the buccal or lingual bony plate of the tooth socket extending no more than 50% of the total depth of the socket.
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non-pregnant women of child-bearing potential.
* Are nonsmokers or former smokers. Current smokers may only be included if they smoke <10 cigarettes per day

Exclusion Criteria:

* Patients who live more than 50 miles from the School of Dentistry, University of Texas Health Science Center at San Antonio
* Patients who do not meet all the inclusion criteria or who will not cooperate with the required follow-up schedule.
* Patients will are mentally incompetent, prisoners, or pregnant.
* Pregnant women or women intending to become pregnant during the study period.
* Smokers who smoke >10 cigarettes per day
* Clinical and/or radiographic determinations which will preclude inclusion in this study are: Active infection other than periodontitis; Inadequate bone dimensions or restorative space for a dental implant; Presence of a disease entity, condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, autoimmune diseases, history of bisphosphonate use or long-term steroid therapy; Positive medical history of endocarditis following oral or dental surgery.
* Sensitivity or allergy to Bacitracin, Gentamicin, Polymyxin B Sulfate, alcohol and/or surfactants

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L. Mealey, DDS, MS, Principal Investigator — UT Health Science Center at San Antonio, School of Dentistry
Locations (1):
- UT Health Science Center at San Antonio, School of Dentistry, San Antonio, Texas, United States

REFERENCES:
- [Derived] Corning PJ, Mealey BL. Ridge preservation following tooth extraction using mineralized freeze-dried bone allograft compared to mineralized solvent-dehydrated bone allograft: A randomized controlled clinical trial. J Periodontol. 2019 Feb;90(2):126-133. doi: 10.1002/JPER.18-0199. Epub 2018 Sep 19. PMID 30161278

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, one subject was withdrawn as a screen failure. This left a total of 43 subjects enrolled to take part in the study
Groups:
- Non-Freeze-Dried Bone Allograft (PUROS): Ridge preservation bone grafting surgery with Non-Freeze-Dried cancellous bone allograft (PUROS)
  PUROS (Ridge Preservation bone grafting surgery): Ridge preservation bone grafting after tooth extraction
- Freeze-Dried Bone Allograft (FDBA): Ridge preservation bone grafting surgery with Freeze-Dried cancellous bone allograft (FDBA)
  FDBA (Ridge Preservation bone grafting surgery): Ridge preservation bone grafting after tooth extraction
Period: Overall Study
Arm/Group | Non-Freeze-Dried Bone Allograft (PUROS) | Freeze-Dried Bone Allograft (FDBA)
Started | 21 | 22
Completed | 18 | 20
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Freeze-Dried Bone Allograft (PUROS) | Freeze-Dried Bone Allograft (FDBA) | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: % Vital Bone Formation (Histological)
Description: histologic determination of % of vital bone formation
Time Frame: 3 months after ridge preservation
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Non-Freeze-Dried Bone Allograft (PUROS) | Freeze-Dried Bone Allograft (FDBA)
Number analyzed (Participants) | 17 | 20
percentage | 27.19 (17.5) | 24.08 (12.49)

2. Secondary Outcome: % Residual Graft Material (Histological)
Description: histologic determination of % of residual bone graft material
Time Frame: 3 months after ridge preservation
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Non-Freeze-Dried Bone Allograft (PUROS) | Freeze-Dried Bone Allograft (FDBA)
Number analyzed (Participants) | 17 | 20
percentage | 23.38 (13.45) | 22.96 (21.04)

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Non-Freeze-Dried Bone Allograft (PUROS) | Freeze-Dried Bone Allograft (FDBA)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Freeze-Dried Bone Allograft (PUROS) (N=21) | Freeze-Dried Bone Allograft (FDBA) (N=22)
Head trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Patient fell at home, head trauma, went into ER, hospitalized for 2 days, MRI, CT scan, obtained medical clearance, follow up in with MD

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT02515058/Prot_SAP_000.pdf